CLINICAL TRIAL: NCT02019927
Title: Evaluation of the Effectiveness and Safety of Transcorneal Electrical Stimulation to Improve Visual Function After Ocular Trauma
Brief Title: Electric Stimulation of the Eye to Improve Vision After Trauma
Acronym: TES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Julia Haller, Evaluation of the Effectiveness of Transcorneal Electrical Stimulation to Improve Visual Function Following Ocular Trauma, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-232
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Non-arteritic Anterior Ischemic Optic Neuropathy (NAION); Trauma; Multiple Sclerosis (MS)
Keywords: NAION; Decreased vision; Eye trauma; TES; Electrical stimulation; Multiple Sclerosis; Optic Neuritis
MeSH Terms: conditions — Wounds and Injuries; Multiple Sclerosis; Optic Neuropathy, Ischemic; Vision Disorders; Eye Injuries; Optic Neuritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Non-arthritic ischemic optic neuropathy (Experimental): Treatment of decreased vision due to NAION with the transcorneal electrical stimulation device (6+ months post-event).
  Interventions: Device: Transcorneal Electrical Stimulation
- Multiple Sclerosis (Experimental): Treatment of decreased vision due to multiple sclerosis with the transcorneal electrical stimulation device (3+ months post visual changes).
  Interventions: Device: Transcorneal Electrical Stimulation
- Ocular Trauma (Experimental): Treatment of decreased vision due to ocular trauma with the transcorneal electrical stimulation device (3+ months post-trauma).
  Interventions: Device: Transcorneal Electrical Stimulation
- Sham - Non-arthritic ischemic optic neuropathy (Sham Comparator): Sham treatment of decreased vision due to NAION with the transcorneal electrical stimulation device (6+ months post-event).
  Interventions: Device: Sham
- Sham - Multiple Sclerosis (Sham Comparator): Sham treatment of decreased vision due to multiple sclerosis with the transcorneal electrical stimulation device (3+ months post visual changes).
  Interventions: Device: Sham
- Sham - Ocular Trauma (Sham Comparator): Sham treatment of decreased vision due to ocular trauma with the transcorneal electrical stimulation device (3+ months post-trauma).
  Interventions: Device: Sham

INTERVENTIONS:
Device: Transcorneal Electrical Stimulation — The clinical trial will investigate whether Transcorneal Electrical Stimulation delivered by the Okuvision Stimulation Set manufactured by Okuvision GmbH, Reutlingen, Germany, is a potentially effective therapy for the restoration and rehabilitation of vision loss as measured by improvements in visual acuity in the following three patient populations: patients with ocular trauma, patients with optic neuritis associated with multiple sclerosis and patients with Non-arteritic Anterior Ischemic Optic Neuropathy.
  Other Names: TES; OkuVision
  Arms: Multiple Sclerosis; Non-arthritic ischemic optic neuropathy; Ocular Trauma
Device: Sham — Sham
  Arms: Sham - Multiple Sclerosis; Sham - Non-arthritic ischemic optic neuropathy; Sham - Ocular Trauma

SUMMARY:
Transcorneal Electrical Stimulation (TES) using the "OkuStim®" device delivers electrical impulses to damaged and/or diseased photoreceptor cells. This electric stimulation of the retina may help to preserve visual acuity and/or the visual field.

DETAILED DESCRIPTION:
The finely detailed, precise anatomy of the retina and optic nerve capture light impulses from the environment through a biochemical process and then transmit these images to the brain via electrical impulses conducted from the inner retina to the optic nerve and ultimately to the occipital cortex.

In the human eye, three types of specialized ganglion cells transmit electrical impulses to the brain. Among these three cell populations are rod and cone cells, which participate in the photo-transduction step of light perception, along with other light sensitive ganglion cells. It is a system whereby the photosensitive pigment rhodopsin (or one of its analogs) rearranges in response to light, and this change in chemical structure fires electrical impulses to the brain which in turn interprets the incoming impulses as a visual image.

Transcorneal Electrical Stimulation (TES) using the "OkuStim®" device delivers electrical impulses to damaged and/or diseased photoreceptor cells. This electric stimulation of the retina may help to preserve VA and/or the visual field.

ELIGIBILITY:
Inclusion Criteria:

* You are 18 years or older.
* You have sustained trauma (more than 3 months before this study) OR been diagnosed with Non-Arteritic Anterior Ischemic Optic Neuropathy (NAION) (more than 6 months before this study) OR been diagnosed with Multiple Sclerosis (MS) and suffered visual loss (more than 3 months before this study).
* You are willing and able to give written informed consent.
* You are able to commit to enrolling in the study during the full time period of up to 6 months.

Exclusion Criteria:

* You have any other significant ophthalmologic disease or condition (such as glaucoma, retinal degeneration, proliferative diabetic retinopathy, +/- six diopters of myopia, retinal detachment, exudative age-related macular degeneration).
* You have amblyopia (lazy eye) in affected eye, previously diagnosed.
* You are participating in any other interventional clinical trial.
* If you are pregnant OR a woman with childbearing potential who is unwilling to use medically acceptable means of birth control for study duration OR woman unwilling to perform a pregnancy test at study entry/screening.
* You are unable to give signed consent due to memory, medical, communication, language, or mental health problems.
* You are less than 18 years old.
* You are unable or unwilling to complete the evaluation or questionnaire.
* Visual acuity better than 20/40
* Inability to detect phosphenes during threshold detection
* You are on seizure medications, or have a history of epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2013-07; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Haller, MD, Principal Investigator — Wills Eye Hospital
Locations (1):
- Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-arteritic Ischemic Optic Neuropathy: Treatment of decreased vision due to NAION with the transcorneal electrical stimulation device (6+ months post-event).
  Transcorneal Electrical Stimulation: The clinical trial will investigate whether Transcorneal Electrical Stimulation delivered by the Okuvision Stimulation Set manufactured by Okuvision GmbH, Reutlingen, Germany, is a potentially effective therapy for the restoration and rehabilitation of vision loss as measured by improvements in visual acuity in the following three patient populations: patients with ocular trauma, patients with optic neuritis associated with multiple sclerosis and patients with Non-arteritic Anterior Ischemic Optic Neuropathy.
- Non-arteritic Ischemic Optic Neuropathy (NAION) Sham: Sham treatment for Non-arteritic ischemic optic neuropathy group
- Multiple Sclerosis Sham: Sham treatment for optic neuritis with Multiple Sclerosis group
- Ocular Trauma Sham: Sham treatment for ocular trauma group
Period: Overall Study
Arm/Group | Non-arteritic Ischemic Optic Neuropathy | Non-arteritic Ischemic Optic Neuropathy (NAION) Sham | Multiple Sclerosis | Multiple Sclerosis Sham | Ocular Trauma | Ocular Trauma Sham
Started | 46 | 23 | 9 | 5 | 10 | 4
Completed | 44 | 19 | 8 | 3 | 7 | 3
Not Completed | 2 | 4 | 1 | 2 | 3 | 1
Not completed — Lost to Follow-up | 2 | 4 | 1 | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Non-arteritic Ischemic Optic Neuropathy Sham: Sham comparator for the Non-arteritic ischemic optic neuropathy group
- Multiple Sclerosis Sham: Sham comparator for the multiple sclerosis group
- Ocular Trauma Sham: Sham comparator for the ocular trauma group
- Total: Total of all reporting groups
Arm/Group | Non-arteritic Ischemic Optic Neuropathy | Non-arteritic Ischemic Optic Neuropathy Sham | Multiple Sclerosis | Multiple Sclerosis Sham | Ocular Trauma | Ocular Trauma Sham | Total
Number analyzed (Participants) | 46 | 23 | 9 | 5 | 10 | 4 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (8.8) | 66 (7.4) | 40.6 (9.7) | 41 (9.2) | 49.2 (14.2) | 45.5 (13.2) | 50.8 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 7 | 3 | 2 | 1 | 37
  Male | 33 | 12 | 2 | 2 | 8 | 3 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 44 | 23 | 9 | 5 | 8 | 4 | 93
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 2 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 2 | 0 | 0 | 6
  White | 43 | 21 | 7 | 3 | 8 | 4 | 86
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 2 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 46 | 23 | 9 | 5 | 10 | 4 | 97

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Effectiveness and Safety of Transcorneal Electrical Stimulation to Improve Visual Acuity
Description: The primary outcomes are change in high-contrast LogMar VA from baseline (week 1) to initial post treatment (week 8). Participants read letters from a chart and receive 1 point for each letter correctly identified. Scores are converted to logMAR scale and analyzed for changes in visual acuity. Improvement in visual acuity is defined as a decrease in logMAR of 0.2 or more.
Time Frame: Change from Baseline (week 1) to 1-week post initial treatment (week 8)
Measure: Mean (95% Confidence Interval); unit: logMAR
Groups:
- Sham - Non-arteritic Ischemic Optic Neuropathy: Sham treatment of decreased vision due to NAION with the transcorneal electrical stimulation device (6+ months post-event).
- Sham - Multiple Sclerosis: Sham treatment of decreased vision due to Multiple Sclerosis
- Sham - Ocular Trauma: Sham treatment of decreased vision due to ocular trauma
Arm/Group | Non-arteritic Ischemic Optic Neuropathy | Sham - Non-arteritic Ischemic Optic Neuropathy | Multiple Sclerosis | Sham - Multiple Sclerosis | Ocular Trauma | Sham - Ocular Trauma
Number analyzed (Participants) | 46 | 23 | 9 | 5 | 10 | 4
logMAR | -0.23 [-0.30 to -0.17] | -0.14 [-0.23 to -0.05] | -0.08 [-0.22 to 0.06] | -0.06 [-0.25 to 0.13] | -0.29 [-0.45 to -0.12] | -0.05 [-0.3 to 0.2]

2. Secondary Outcome: Intra-Ocular Pressure (IOP)
Description: Measured by Applanation (Galdmann) Tonometry method
Time Frame: Change from Baseline (week 1) to 1-week post initial treatment (week 8)
Measure: Mean (95% Confidence Interval); unit: mmHg
Groups:
- Sham - Non-arteritic Ischemic Optic Neuropathy (NAION): Sham treatment of decreased vision due to NAION
- Sham - Multiple Sclerosis (MS): Sham treatment of decreased vision due to MS
Arm/Group | Non-arteritic Ischemic Optic Neuropathy | Sham - Non-arteritic Ischemic Optic Neuropathy (NAION) | Multiple Sclerosis | Sham - Multiple Sclerosis (MS) | Ocular Trauma | Sham - Ocular Trauma
Number analyzed (Participants) | 41 | 21 | 6 | 5 | 8 | 2
mmHg | -0.32 [-0.99 to 0.34] | -1.13 [-2.06 to -0.20] | -0.27 [-3.26 to 2.72] | 0.52 [-2.77 to 3.81] | 0.52 [-1.57 to 2.6] | -0.57 [-4.78 to 3.63]

3. Secondary Outcome: Visual Field Mean Deviation
Description: The Humphrey 24-2 Swedish Interactive Threshold Algorithm Standard perimeter was used to test visual field. Reported values are a change from baseline to 1-week post initial treatment.
Time Frame: Change from Baseline (week 1) to 1 - week post initial treatment (week 8)
Measure: Mean (95% Confidence Interval); unit: Decibels (dB)
Groups:
- Sham - NAION: Sham treatment of decreased vision due to NAION
Arm/Group | Non-arteritic Ischemic Optic Neuropathy | Sham - NAION | Multiple Sclerosis | Sham - Multiple Sclerosis | Ocular Trauma | Sham - Ocular Trauma
Number analyzed (Participants) | 44 | 23 | 9 | 5 | 9 | 4
Decibels (dB) | 1.49 [0.72 to 2.25] | 2.09 [1.03 to 3.15] | 1.31 [-0.94 to 3.55] | 0.96 [-2.21 to 4.13] | 1.70 [0.23 to 3.18] | 0.25 [-1.98 to 2.48]

4. Secondary Outcome: Ocular Coherent Tomography, Retinal Nerve Fiber Layer Thickness in Superior Quadrant
Description: Assessed the change in thickness of the retinal nerve fiber layer 1-week post treatment compared to baseline
Time Frame: Change from Baseline (week 1) to 1 - week post initial treatment (week 8)
Measure: Mean (95% Confidence Interval); unit: um
Arm/Group | Non-arteritic Ischemic Optic Neuropathy | Sham - NAION | Multiple Sclerosis | Sham - Multiple Sclerosis | Ocular Trauma | Sham - Ocular Trauma
Number analyzed (Participants) | 42 | 21 | 9 | 5 | 9 | 4
um | -0.70 [-9.92 to 8.52] | 12.41 [-0.66 to 25.47] | -3.80 [-12.97 to 5.37] | -5.97 [-18.86 to 6.92] | 0.37 [-2.13 to 2.87] | 1.42 [-2.33 to 5.17]

5. Secondary Outcome: Ocular Coherent Tomography, Retinal Nerve Fiber Layer Thickness in Nasal Quadrant
Description: Assessed the change in thickness of the retinal nerve fiber layer 1-week post treatment compared to baseline
Time Frame: Change from Baseline (week 1) to 1 - week post initial treatment (week 8)
Measure: Mean (95% Confidence Interval); unit: um
Arm/Group | Non-arteritic Ischemic Optic Neuropathy | Sham - NAION | Multiple Sclerosis | Sham - Multiple Sclerosis | Ocular Trauma | Sham - Ocular Trauma
Number analyzed (Participants) | 42 | 21 | 9 | 5 | 9 | 4
um | -0.48 [-2.64 to 1.69] | -1.24 [-4.30 to 1.82] | -3.60 [-9.33 to 2.12] | 0.28 [-7.69 to 8.26] | 0.49 [-1.66 to 2.65] | -1.36 [-4.59 to 1.88]

6. Secondary Outcome: Ocular Coherent Tomography, Retinal Nerve Fiber Layer Thickness in Inferior Quadrant
Description: Assessed the change in thickness of the retinal nerve fiber layer 1-week post treatment compared to baseline
Time Frame: Change from Baseline (week 1) to 1 - week post initial treatment (week 8)
Measure: Mean (95% Confidence Interval); unit: um
Arm/Group | Non-arteritic Ischemic Optic Neuropathy | Sham - NAION | Multiple Sclerosis | Sham - Multiple Sclerosis | Ocular Trauma | Sham - Ocular Trauma
Number analyzed (Participants) | 42 | 21 | 9 | 5 | 9 | 4
um | -0.04 [-1.28 to 1.21] | -0.64 [-2.40 to 1.12] | -2.37 [-6.94 to 2.19] | 1.07 [-5.23 to 7.37] | 0.57 [-2.03 to 3.16] | -1.53 [-5.51 to 2.46]

7. Secondary Outcome: Ocular Coherent Tomography, Retinal Nerve Fiber Layer Thickness in Temporal Quadrant
Description: Assessed the change in thickness of the retinal nerve fiber layer 1-week post treatment compared to baseline
Time Frame: Change from Baseline (week 1) to 1 - week post initial treatment (week 8)
Measure: Mean (95% Confidence Interval); unit: um
Arm/Group | Non-arteritic Ischemic Optic Neuropathy | Sham - NAION | Multiple Sclerosis | Sham - Multiple Sclerosis | Ocular Trauma | Sham - Ocular Trauma
Number analyzed (Participants) | 42 | 21 | 9 | 5 | 9 | 4
um | 2.15 [-2.43 to 6.73] | -0.64 [-2.40 to 1.12] | -0.49 [-1.62 to 0.64] | 1.07 [-5.23 to 7.37] | -0.35 [-1.71 to 1.00] | -1.53 [-5.51 to 2.46]

8. Secondary Outcome: Ocular Coherent Tomography, Retinal Nerve Fiber Layer Thickness in Center Quadrant
Description: Assessed the change in thickness of the retinal nerve fiber layer 1-week post treatment compared to baseline
Time Frame: Change from Baseline (week 1) to 1 - week post initial treatment (week 8)
Measure: Mean (95% Confidence Interval); unit: um
Arm/Group | Non-arteritic Ischemic Optic Neuropathy | Sham - NAION | Multiple Sclerosis | Sham - Multiple Sclerosis | Ocular Trauma | Sham - Ocular Trauma
Number analyzed (Participants) | 37 | 22 | 8 | 5 | 7 | 4
um | -0.07 [-4.43 to 4.23] | 3.89 [-1.79 to 9.55] | -2.83 [-7.63 to 1.97] | -1.07 [-7.34 to 5.19] | -0.62 [-2.14 to 0.91] | -0.42 [-2.50 to 1.66]

9. Secondary Outcome: National Eye Institute's Visual Functioning Questionnaire - 25
Description: Test to measure Unweighted of scores within test ranging from 0-100 with higher scores meaning better outcome
Time Frame: Change from Baseline to 1 - week post initial treatment
Measure: Mean (95% Confidence Interval); unit: score on a scale - change from baseline
Arm/Group | Non-arteritic Ischemic Optic Neuropathy | Sham - NAION | Multiple Sclerosis | Sham - Multiple Sclerosis | Ocular Trauma | Sham - Ocular Trauma
Number analyzed (Participants) | 45 | 23 | 9 | 5 | 9 | 4
score on a scale - change from baseline | -0.59 [-2.41 to 1.24] | 0.16 [-2.40 to 2.72] | 4.59 [-2.55 to 11.73] | 4.57 [-5.08 to 14.22] | 3.64 [-1.40 to 8.67] | 5.27 [-2.51 to 13.04]

10. Secondary Outcome: Symbol Digit Modality Testing
Description: Scores range from 0-110 with higher scores meaning better visual information processing speed
Time Frame: Change from Baseline to 1 - week post initial treatment
Measure: Mean (95% Confidence Interval); unit: score on a scale - change from baseline
Arm/Group | Non-arteritic Ischemic Optic Neuropathy | Sham - NAION | Multiple Sclerosis | Sham - Multiple Sclerosis | Ocular Trauma | Sham - Ocular Trauma
Number analyzed (Participants) | 30 | 14 | 7 | 5 | 7 | 3
score on a scale - change from baseline | -0.03 [-2.42 to 2.37] | -0.01 [-3.52 to 3.50] | 2.98 [-1.70 to 7.66] | -0.77 [-6.48 to 4.94] | 4.08 [-2.19 to 10.36] | 6.14 [-3.58 to 15.86]

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Sham - Non-arteritic Ischemic Optic Neuropathy: Sham treatment of decreased vision due to NAION
Arm/Group | Non-arteritic Ischemic Optic Neuropathy | Sham - Non-arteritic Ischemic Optic Neuropathy | Multiple Sclerosis | Sham - Multiple Sclerosis | Ocular Trauma | Sham - Ocular Trauma
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/23 | 0/9 | 0/5 | 0/9 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/23 | 0/9 | 0/5 | 0/9 | 0/4
Other Adverse Events (participants affected / at risk) | 15/45 | 0/23 | 3/9 | 0/5 | 5/9 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-arteritic Ischemic Optic Neuropathy (N=45) | Sham - Non-arteritic Ischemic Optic Neuropathy (N=23) | Multiple Sclerosis (N=9) | Sham - Multiple Sclerosis (N=5) | Ocular Trauma (N=9) | Sham - Ocular Trauma (N=4)
Minor ocular surface irritation (Eye disorders) | 15 (15) | 0 (0) | 3 (3) | 0 (0) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT02019927/Prot_SAP_000.pdf